CLINICAL TRIAL: NCT03236727
Title: SSEP Fluctuations Due to Dexmedetomidine During Posterior Spine Fusion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: George Papanicolaou Hospital (Other)
Responsible Party: Principal Investigator, Asouhidou Irene, Assistant Professor, George Papanicolaou Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: GeorgePHT
Record Dates: First submitted 2017-07-25; First posted 2017-08-02 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Spinal Fusion
Keywords: Dexmedetomidine, spinal fusion, SSEP
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Data of SSEPs (amplitude and latency) before dexmedetomidine infusion.
- Dexmedetomidine (Active Comparator): Data of SSEPs (amplitude and latency) after dexmedetomidine infusion.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Changes of both amplitude and latency of SSEPs during dexmedetomidine infusion.
  Other Names: Control-no dexmedetomidine
  Arms: Dexmedetomidine

SUMMARY:
Intravenous anesthetic agents as far as inhaled agents produce a dose depended increase in latency and decrease in amplitude of SomatoSensory Evoked Potential (SSEP). Dexmetedomidine, a highly selective a2 adrenergic agonist, not only minimizes the anesthetic agents but also the opioids, reducing the analgesic demands. The effect of dexmedetomidine on SSEP has not been elucidated. We aimed to investigate alterations on somatosensory SSEP in adults during posterior spinal fusion surgery before and after Dexmedetomidine administration.

DETAILED DESCRIPTION:
Patients 18-75 years old, ASA (physical status classification system) I-III, scheduled for elective posterior spinal fusion surgery were enrolled in this prospective study. After induction in anesthesia, it was applied SSEP monitoring and a baseline test was performed after 15min (in order to wash out the propofol used for induction). Infusion of Dexmedetomidine was started at a bolus dose of 1mcg/Kg following by 0.7mcg/Kg. Bispectral Index (BIS) monitored the depth of anesthesia and an adequate level (40-50) of anesthesia was maintained by sevoflurane. SSEP were recorded intraoperatively from the tibial nerve (P37) and data were analyzed over that period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA physical status 1-3

Exclusion Criteria:

* Patients with ASA physical status >3,
* Body Mass Index (BMI) over 30,
* indication for rapid sequence induction,
* any contraindication for receiving b-blocker,
* Glasgow Coma Scale (GCS) <13,
* history of drug abuse,
* neurologic deficit or preoperatively foreseen delayed extubation,
* preoperative heart rate<45.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
SSEPs | 10 min after starting infusion of dexmedetomidine
  measurement of SSEPs parameters regarding the baseline.